CLINICAL TRIAL: NCT01600846
Title: Delivery of Pharmacogenetic Testing in a Primary Care Setting
Brief Title: Pharmacogenetic Testing in Primary Care
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00031122; 2R01GM081416-04 (NIH)
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2014-08

CONDITIONS: Pharmacogenetic Testing
Keywords: Pharmacogenetic testing; pharmacokinetics; Pharmacogenomics; genetics; pharmacy; drug response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to further integrate pharmacogenetic (PGx) testing into clinical practice by educating physicians about pharmacogenetics and offering testing to their patients. Pharmacogenetic testing may help physicians choose the best drug and dosage for their patients which can reduce side effects, increase effectiveness, and improve patient adherence.

Two clinics will be involved. One clinic will have a pharmacist on-site as a resource to physicians and to advise what patients may benefit from PGx testing; the other clinic will have a pharmacist on call.

Patient and physician perspectives about PGx testing and their utilization will be examined via surveys.

The investigators hypothesize that with education about PGx testing, more physicians will utilize testing.

DETAILED DESCRIPTION:
This study aims to assess two delivery models of PGx testing (physician-initiated and pharmacist-initiated) for commonly prescribed drugs in primary care practices and evaluate the delivery of testing from three perspectives: physician, patient, and practice setting. We hypothesize that greater utilization will be influenced by increased physician knowledge and awareness of drugs with PGx testing, comfort in discussing PGx testing with patients and applying results to therapeutic decision-making and positive attitudes towards the testing process. We hypothesize that the pharmacist-initiated approach will result in the most effective use and rapid uptake of PGx testing given the hands-on educational approach with the pharmacist providing expert guidance. We also hypothesize that having a pharmacist with PGx testing expertise as part of the medical team will result in greater physician comfort with test ordering and application of results as compared with the physician-initiated model. In addition, an economic analysis will be conducted to evaluate and compare the costs of each model.

We will also examine patient perspectives about PGx testing and their utilization of test results. We hypothesize that patients who have experienced adverse responses or a poor drug outcome (no response) in the past, are taking chronic medications, and those who are older will be more likely to consent to PGx testing. We hypothesize that patients' increased awareness about their genetic predisposition to adverse responses will result in greater discussion with prescribing physicians and pharmacists about the PGx results when new treatments are prescribed, with greater attention to adverse effects of new drugs and potentially greater medication compliance.

We will implement and evaluate two delivery models of PGx testing into primary care practices: physician-initiated testing and pharmacist-initiated testing. Each practice will be provided an educational intervention and will be surveyed prior to the seminar and following the intervention period to assess primary care practitioner (PCP) knowledge and attitudes about PGx testing. These surveys will take about 10-15 minutes to complete and will be available through an online system like SurveyMonkey.

In the pharmacist-initiated group, a pharmacist based within the practice will identify prescribed drugs with available PGx testing through chart review and provide specific information and recommendations about PGx testing to the ordering physician. In the physician-initiated group, physicians will order testing as they deem necessary, but will also have on-call pharmacist support to consult.

Patients who are offered PGx testing will also be surveyed: once after deciding whether or not to pursue PGx testing and then, if they consent to testing, after they receive their test results. These surveys will take about 10-15 minutes to complete and will be on paper (pretest) and online through a system like SurveyMonkey (post-test). The pretest survey will have 3 sections: demographics, perceived risks and benefits of PGx testing, and satisfaction with test results. The post-test will assess information-seeking behavior, medication adherence, and knowledge of adverse drug reactions.

Chart reviews will be conducted throughout the study to collect various data-points. All extracted data-points will be coded; the key will be stored in a separate file to minimize any breach of privacy. In summary, the medical records of patients scheduled to be seen at either clinic during the first or second phase of the study (see Figure 1) will be reviewed to identify those patients that were prescribed a drug from Table 1. A post-intervention (the third and final phase of the study) chart review will be conducted to monitor the number of new prescriptions for drugs listed in Table 1, the frequency with which PGx testing is ordered, by which physicians, and for which drugs.

We will conduct chart reviews at the end of each phase of the study (pre-intervention period, intervention period, and post intervention period) of patients prescribed targeted medications. No HIPAA (Health Insurance Portability and Accountability Act) identifiers will be recorded.

All PCPs practicing at the two clinics involved in the study are eligible to participate. All physicians who participate in the educational intervention in either arm will be invited to participate in the pre and post-intervention surveys.

The patient survey population will include patients who were offered and consented or declined testing. All patients 18 years and older who were prescribed a drug for which PGx testing is available and offered a PGx test by their physician during the intervention period will be asked to participate in the initial survey. Patients must be English-speaking and able to complete the survey without assistance.

Chart review will include all patients who were scheduled an appointment at either of the clinics within the designed study period. Data abstracted (full chart review) will be limited to those patients who were prescribed a target drug during the designated period.

ELIGIBILITY:
Inclusion Criteria:

* must be a patient or physician at one of the participating clinics
* patients must be prescribed a medication that has PGx testing available
* 18 years of age or older
* English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physician population will be physicians practicing at the two clinics part of Duke University Medical Center Patient population will be patients who receive primary care at one of the two participating clinics.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Use of PGx testing | 6 months, 12 months

SECONDARY OUTCOMES:
Number of adverse drug reactions | 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Haga, PhD, Principal Investigator — Duke Unviersity Medical Center
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States